CLINICAL TRIAL: NCT01937832
Title: A Phase III Study to Evaluate the Efficacy and Safety of Faropenem in the Treatment of Adult Community-acquired Bacterial Pneumonia
Brief Title: A Phase III Study of Faropenem in the Treatment of Adult Community-acquired Bacterial Pneumonia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTTQ04104-3-CTF
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — fropenem; Ertapenem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ertapenem (Active Comparator)
  Interventions: Drug: Ertapenem
- Faropenem (Experimental)
  Interventions: Drug: Faropenem

INTERVENTIONS:
Drug: Faropenem — dosage form: Injection dosage:1200 mg frequency: Three times a day
  Arms: Faropenem
Drug: Ertapenem — dosage form: Injection dosage:1000 mg frequency: once a day
  Arms: Ertapenem

SUMMARY:
The purpose of this study is to evaluate the safety and Efficacy of Faropenem in community-acquired pneumonia (CAP) subjects

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between18~73 years, either male or female
2. Patients requiring hospitalization or emergency room observation, and the need to receive intravenous antibiotic treatment
3. Women of childbearing age having negative pregnancy test at the time of enrollment and agreeing to take effective contraceptive measures from the delivery to 7 ~14 days after stopping .(for example: oral contraception, injectable contraception, or implant contraception , spermicides and condoms, or IUDs).
4. Comply with the following clinical, radiological and microbiological criteria of Community-Acquired Pneumonia(CAP)
5. Patients had used ineffective systemic antimicrobial drugs before enrollment or had effective antimicrobial drugs within 72h before enrollment, used <24h
6. Informed consent granted

Exclusion Criteria:

1. Patients with atypical pneumonia infected by the Mycoplasma pneumoniae, Chlamydia pneumoniae, Legionella pneumophila bacteria;
2. Patients infected by pathogens MRSA, Pseudomonas aeruginosa or Acinetobacter baumannii;
3. Viral pneumonia;
4. Aspiration pneumonia;
5. Hospital-acquired pneumonia, including ventilator-associated pneumonia;
6. Patients with Severe pneumonia who meet one primary criterion or three secondary criteria (See Appendix);
7. Patients with a rapid progressive or end-stage disease, and can not survive until the end of the study period by antibiotic treatment;
8. Patients with bronchial obstruction or a history of obstructive pneumonia (not including chronic obstructive pulmonary disease);
9. Suffering from any of the following diseases: active tuberculosis, bronchiectasis, lung abscess, lung cancer, non-infectious interstitial lung disease, pulmonary edema, atelectasis, pulmonary embolism, pulmonary eosinophil infiltration disease and pulmonary vasculitis;
10. Infections acquired from hospitals, nursing homes or other long-term care facilities, or patients hospitalized within 14 days prior to enrollment ;
11. Allergic to penem and carbapenem antibiotic;
12. Pregnancy or lactation in women;
13. Patients with uncontrolled psychiatric history or those at risk of suicide two years prior to enrollment;
14. A history of epilepsy or other central nervous system disorders in patients;
15. Patients with Renal dysfunction, screening serum creatinine values above the upper limit of normal 10%;
16. The Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is 3 times the upper limit of the reference value, or total bilirubin beyond the upper limit of the normal range by 10% ;
17. Serious diseases that affecting the immune system, such as: a human immunodeficiency virus (HIV) infection history, or CD4 + T-lymphocyte count <200/200/mm3, or Neutrophilic granulocytopenia (neutrophil count <1500/mm3), or hematologic malignancies or solid organ or splenectomy, etc;
18. Patients who are taking steroid medications, at least 20mg daily dose of prednisone(or equivalent doses of other glucocorticoids);
19. Patients who are accepting chemotherapy drug therapy or anti-cancer therapy, or plan to accept such treatment during the trial six months prior to enrollment;
20. Alcohol or illicit drug abuse history;
21. Patients who have accepted any other experimental drugs within 3 months prior to enrollment;
22. more than 500ml blood donation within 3 months prior to enrollment;
23. Patients who have participated in this clinical trial ever before;
24. Combined use of other antibacterial drugs in patients;
25. Patients are diagnosed to have potential increased risks, or there may be interference with clinical trials;

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Per subject clinical cure rate | 7-14 days

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Taihe Hospital in Shiyan City, Shiyan, Hubei
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Huashan Hospital ,Fudan University, Shanghai
  - The Second Hospital of Tianjin Medical University, Tianjin